CLINICAL TRIAL: NCT02407080
Title: Open Label Phase I Study of Single Agent Oral RG7388 in Patients With Polycythemia Vera and Essential Thrombocythemia (With Pilot Feasibility Study in Combination With Pegylated Interferon Alfa 2a for Patients Who do Not Respond to the Single Agent at Each Dose Level)
Brief Title: Open Label Study of Single Agent Oral RG7388 in Patients With Polycythemia Vera and Essential Thrombocythemia
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: John Mascarenhas (Other)
Collaborators: Roche Pharma AG (Industry); The Leukemia and Lymphoma Society (Other)
Responsible Party: Sponsor-Investigator, John Mascarenhas, Associate Professor, Icahn School of Medicine at Mount Sinai
Organization: Icahn School of Medicine at Mount Sinai (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GCO 12-0481-1001; MPD-RC 115 (Other: Myeloproliferative Disorders-Research Consortium); GCO 14-1919 (Other: Icahn School of Medicine at Mount Sinai)
Record Dates: First submitted 2015-03-24; First posted 2015-04-02 (Estimated); Last update posted 2019-09-12 (Actual); Status verified 2019-09

CONDITIONS: Polycythemia Vera; Essential Thrombocythemia
MeSH Terms: conditions — Polycythemia Vera; Thrombocythemia, Essential | interventions — RG7388; peginterferon alfa-2a

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- RG7388 (Experimental): Part A: RG7388 as a single agent; given at a starting dose of 100 mg each day for five days for the first cycle which will be 56 days.
  Part B: combination of RG7388 and Pegasys if subject does not achieve at least a PR by the end of 3 cycles of single agent RG7388
  Interventions: Drug: RG7388; Drug: Pegasys

INTERVENTIONS:
Drug: RG7388 — RG7388 is supplied as film-coated tablets at dosage strengths of 50 mg, 200 mg, 300mg and 400 mg.
Drug: Pegasys — PEGASYS is supplied as a clear, sterile solution for subcutaneous (SQ) injection available in prefilled syringes. weekly doses at 45ug subcutaneously
  Other Names: pegylated interferon alfa-2a

SUMMARY:
This research looks at two conditions, Essential Thrombocythemia (ET) and Polycythemia Vera (PV). ET causes people to produce too many blood cells called platelets and PV causes too many platelets and red blood cells to be made. Platelets are particles which circulate in the blood stream and normally prevent bleeding and bruising. Having too many platelets in the blood increases the risk of developing blood clots, which can result in life threatening events like heart attacks and strokes. When the number of red blood cells is increased in PV this will slow the speed of blood flow in the body and increase the risk of developing blood clots.

The purpose of Part A of this study is to test the safety and tolerability of drug RG7388 patients and identify the recommended phase II dose in a single agent dose escalation study. The investigators want to find out what effects, good and/or bad it has on the disease.

The purpose of Part B of this study is to test the safety and tolerability of the combination of RG7388 and Pegylated Interferon Alfa-2a or Pegasys in PV/ET patients from Part A who did not achieve at least a partial response by the end of three cycles of single agent RG7388.

Essential Thrombocythemia (ET) and Polycythemia Vera (PV) have been difficult diseases to treat. RG7388 is a selective inhibitor of the p53-MDM2 binding that frees p53 from negative control and activates the p53 pathway in cancer cells, leading to cell cycle arrest and apoptosis in vitro and in vivo. It has been used to treat solid tumors and Acute Myelogenous Leukemia (AML) in clinical trials. Pegasys is a drug that is the standard of care for patients who have Chronic Hepatitis B (CHB).

RG7388 is a drug that is not yet approved by the Federal Drug Administration (FDA) for the treatment of patients with essential thrombocythemia or polycythemia vera. Pegasys is a drug that is approved by the FDA for the treatment of CHB. The use of RG7388 alone and in combination with Pegasys is experimental.

DETAILED DESCRIPTION:
The Philadelphia chromosome-negative chronic myeloproliferative neoplasms (MPNs) are a group of hematopoietic stem cell malignancies that include polycythemia vera (PV), essential thrombocythemia (ET), and primary myelofibrosis (PMF). PV and ET can evolve into myelofibrosis, termed post PV/ET MF. ET, PV and PMF have variable tendencies to transform to blast phase disease with a dismal prognosis. JAK2V617F is a point activating mutation resulting in the constitutive activity of the JAK-STAT pathway within hematopoietic cells in approximately 96%, 50%, and 50% of patients with PV, ET, and MF, respectively.

Polycythemia Vera is characterized by an absolute increase in red cell mass. Patients with PV have a median survival if untreated of approximately 18 months from the time of diagnosis and treated of approximately 18 years. PV-related symptoms include headache, weakness, dizziness, epigastric distress, and pruritus. PV-related signs include hypertension, gout, left upper abdominal quadrant pain, high hematocrit, leukocytosis, and thrombocytosis. Major causes of reduced survival include thrombosis (29%), bleeding (7%), evolution to myelofibrosis (3%), transformation to acute leukemia (23%), and solid tumors (16%). PV patients are stratified for risk of thrombosis by age >60 and history of prior thrombotic events. Therapy for low risk PV includes low dose aspirin and therapeutic phlebotomy to maintain a hematocrit <45% in a man and 42% in a woman. Cardiovascular risk factor modification such as weight loss, control of hypertension and hypercholesterolemia, and smoking cessation are also important adjunctive approaches to all patients with PV. High risk patients are also treated with cytoreductive therapy in the form of hydroxyurea to further reduce the risk of thrombotic complications.

Essential Thrombocythemia is characterized by persistent isolated thrombocytosis and tendency for arterial and venous thrombosis. A similar pattern of symptoms as noted above with PV are also seen in patients with ET. The median survival of patients with ET is similar to that of age and sex matched cohort and in some patients is limited by thrombotic complications (22%), evolution to MF (10%), and acute leukemia (2%) (Barbui. J Clin Oncol. 2011; 29(23):3179). Risk stratification for occurrence of thrombosis is based on age >60 years and/or history of thrombosis. Additionally, cardiovascular risk factors and persistent thrombocytosis >1.5 x 109/L are believed to influence thrombotic risk and leukemic transformation has been shown to be associated with anemia, older age, and leukocytosis. JAK2V617F is present in approximately 50% of cases and helps establish a diagnosis of a clonal thrombocytosis, and has been shown in some studies to predict for a higher risk of thrombosis and potential for transformation to PV. Management is aimed at reducing thrombotic risk with the use of low dose aspirin in low risk patients (no risk factors) and cytoreductive therapy in high risk patients (at least one risk factor). Hydroxyurea, anagrelide, and interferon (IFN) have all been used to maintain a platelet count below 400 x 109/L in patients with a history of thrombosis (secondary prophylaxis). Currently, hydroxyurea is considered standard of care for high risk ET patients based on the results of the PT-1 study which demonstrated superiority of hydroxyurea over anagrelide in arterial thrombosis risk reduction and worsening marrow reticulin fibrosis in patients receiving anagrelide (Harrison N Engl J Med. 2005;353(1):33). Hydroxyurea is associated with a risk of oral and skin ulcers, rash, and unacceptable myelosuppression that can sometimes limit use in patients with ET/PV. Additionally, some patients are unable to achieve adequate control of blood counts at doses below 2000 mg/daily and this has been termed "resistance". Importantly, although a theoretical concern of leukemogenic potential of hydroxyurea exists, based on the mechanism of action of this chemotherapeutic agent, there are no definitive prospective studies clearly documenting an increased risk of leukemic transformation.

More recently, a renewed interest in interferon-α for the treatment of PV as an alternative therapeutic approach has led to the evaluation of pegylated interferon-α 2a (Pegasys, Roche) in several phase II studies. Pegasys has an improved toxicity profile over intron-a and can be self-administered by the patient on a weekly basis. Currently, Pegasys is being evaluated in two large international trials within the myeloproliferative disorder research consortium (MPD-RC). The MPD-RC 111 study is a phase II study intended to evaluate the response by European LeukemiaNet (ELN) criteria in patients with high risk ET/PV who are intolerant or resistant to hydroxyurea therapy treated with Pegasys. In addition, patients with documented JAK2V617F and splanchnic vein thrombosis are also eligible for this clinical trial. MPD-RC 112 is a phase III study for newly diagnosed high risk PV/ET patients in which patients are randomized to either Pegasys or hydroxyurea with a primary endpoint of response rate comparison between the two treatment arms.

The use of intron-a (rIFN-α) and Pegasys has been extensively studied in patients with PV and reported rates of discontinuation in the first year of therapy range from 14-40%. Objective hematologic responses are seen in approximately 80% of treated patients and achievement in complete phlebotomy free state in 60% of PV patients. Trials of Pegasys in the treatment of PV have further demonstrated major molecular responses of 19% and complete eradication of JAK2V617F in 14-24% of patients. Although hematologic remission can often be achieved within months of starting rIFN-α treatment, molecular responses require longer term administration and are rarely seen before completion of 12 months of therapy. Additionally, sustained molecular remissions have been documented in patients that have discontinued therapy for up to 30 months of follow up. In a retrospective review of 118 MPN patients receiving Pegasys throughout multiple MPN centers included 55 PV patients with an ORR of 87% (54% CR, 33% PR) by ELN criteria [21]. In this review, the most common non-hematologic toxicities were Grade 1-3 fatigue in 24 patients (20%), Grade 1 liver function test (LFT) elevation in 7 (6%), and Grade 1-2 skin/allergic reaction in 6 (5%). Adverse effects leading to discontinuation were primarily non-hematologic, although one patient (<1%) discontinued Pegasys therapy due to Grade 2 anemia.

Although the biological mechanism of recombinant IFN in the treatment of PV is not completely understood, evidence to suggest promotion of immunoregulatory cell function, inhibition of angiogenesis, induction of pro-apoptotic gene expression, alteration of the bone marrow microenvironment, suppression of hematopoietic progenitor cells, and increase cycling of hematopoietic stem cells (HSC) has been reported.

In the last several years, oral small molecule tyrosine kinase inhibitors of JAK2 have been tested in both pre-clinical and clinical trials of patients with MPNs including PV/ET. These agents have demonstrated remarkable responses in terms of reduction in splenomegaly and correction of leukocytosis, erythrocytosis, and thrombocytosis. However, mature follow up of PV patients treated with JAK2 inhibitors evaluating reduction in thrombotic risk and evolution to MF is not known. Currently, Ruxolitinib (Jakafi) is being evaluated in a phase III study in patients with high risk PV that are refractory/intolerant to hydroxyurea [Response trial: NCT01243944].

The tumor suppressor p53 plays an integral role in the regulation of the cell cycle, apoptosis, DNA repair, and senescence. Fifty percent of cancers are found to have inactivating mutations of p53. Although, inactivating mutations of p53 are uncommon in the chronic phases of MPNs, they increase in frequency in the blast phase of MPNs. The p53 pathway can also be down-regulated in MPN cells that express wild-type p53 through alternative pathways. Over-expression of the ubiquitin ligase murine double minute 2 (MDM2; HDM2 in humans) is a regulator of wild type p53 through a variety of different mechanisms. MDM2 1) promotes proteosomal degradation and 2) inhibits p53 transcription, and 3) inhibits transactivation 4) facilitates export from the nucleus. Inhibition of MDM2 is expected to release the negative regulation of p53 and ultimately promote tumor suppressor function. MDM2 overexpression can be a consequence of gene amplification, increased transcription, and increased translation. It has previously been shown that in primary hematopoietic cells from patients with JAK2V617F PV, reduced expression of p53 is a result of increased La autoantigen expression leading to increased translation of MDM2. It would appear that JAK2V617F induces this ribonucleoprotein and furthermore, La protein expression can be down-regulated by in vitro JAK2 inhibitor treatment. Lu et al demonstrated increased MDM2 expression and reduced p53 levels in JAK2V617F-positive PV CD34+ cells. The physical structure and interaction of p53 and MDM2 is known and has allowed for the development of small molecule inhibitors of MDM2-p53 interaction. Nutlin-3, a small molecule antagonist of MDM2, was shown to inhibit the proliferation of PV CD34+ cells through increased p53 mediated apoptosis. Moreover, in vitro combination of low doses of Pegasys with nutlin-3 resulted in selective and significant inhibition of JAK2V67F-positive CD34+ PV colony formation compared to normal colony formation. Thus, MDM2 appears to be a novel therapeutic target in JAK2V617F-positive PV and ultimately may prove to be most effective when used in combination with Pegasys.

RG7388 is an MDM2-p53 binding cell cycle inhibitor (antiproliferative) and is expected to be myelosuppressive at sufficiently high doses. Nonclinical safety findings with RG7388 that may have potential clinical relevance include thrombocytopenia and neutropenia, as well as general pancytopenia, and effects on liver function parameters.

Clinical experience to date suggests a dose relationship for RG7388 and gastrointestinal AEs with increased incidence of nausea, vomiting, and diarrhea at higher dose levels; gastrointestinal prophylaxis with anti-emetics is recommended. Cytopenias, manifesting as thrombocytopenia and neutropenia, occurring at higher dose levels appear to be related to exposure.

Iancu-Rubin et al have investigated the biological effect of RG7112 (first generation MDM2 inhibitor) induced p53-MDM2 disruption on megakaryopoiesis and platelet production in order to better elucidate the mechanism of treatment associated thrombocytopenia (ASH 2012). Bone marrow derived CD34+ cells exposed to RG7112 for 7 days generated fewer viable cells, fewer CFU-MK colonies as compared to untreated cells. Based on these findings, it would appear that RG7112 impacts megakaryopoiesis by two potential mechanisms: 1) Impairing the ability of CD34+ cells to generate MK precursors due to increased apoptosis; 2) Limiting DNA synthesis and polyploidization during the late stages of MK development due to pharmacological activation of p53. A combination of these two effects may provide an explanation for thrombocytopenia observed in patients receiving this drug and suggests that p53 plays an important role in normal human thrombocytopoiesis.

Study NP27872 is a multi-center, open-label, first-in-human, Phase I dose-escalation study of single agent RG7388, a small molecule MDM2 antagonist, administered orally in patients with advanced malignancies except leukemia. The first patient received RG7388 on 15 November 2011. As of 13 September 2012, 51 patients have been enrolled in the study.

Evaluable PK data is available for 22 patients in Study NP27872. There has been no evidence of significant accumulation (defined as a mean ratio of area under the curve [AUC]τ [on Day 15 or 5] to AUCinf [on Day 1] > 2) observed in the study thus far, except for one patient who exhibited a long half-life (t½) and consequently had an accumulated drug exposure that increased 5-fold from Day 1 to Day 5. This was possibly due to concomitant controlled-release oxycodone, as opioids are known to cause delayed gastric emptying and decreased intestinal motility. In addition, data from the study demonstrate an approximately linear dose-exposure (Day 1 maximum plasma concentration [Cmax]) relationship in RG7388 with moderately high inter-patient variability without an absorption plateau to date.

Macrophage inhibitory cytokine (MIC-1, a secreted protein that is strongly induced by activated p53) serum levels has been used to assess pharmacodynamic (PD) effects in this Phase I study. Analysis of patients on 100 to 800 mg/day of RG7388 showed that the minimum level for p53 induction occurs at a dose of 100 mg/day or a corresponding plasma level of 500 ng/mL of RG7388. Preliminary analysis of PK and safety data showed that there is an apparent PK/PD relationship between an AUC per cycle and Cycle 1 platelet nadir.

At the data cutoff of 13 September 2012, 51 patients with advanced malignancies had received R05503781 in Study NP27872. Fifty patients experienced at least 1 adverse event (AE) and 11 patients experienced at least 1 serious adverse event (SAE).

Thirteen SAEs in patients (white blood cell count decreased, platelet count decreased, 2 cases of neutrophil count decreased, febrile neutropenia, 5 cases of thrombocytopenia, 2 cases of neutropenia, and diarrhea) were considered by the investigator to be probably related to study treatment; 4 SAEs (2 cases of febrile neutropenia, urinary tract infection, and anemia) were considered possibly related; 1 SAE (lung infection) was considered remotely related; and the other 6 SAEs (infection, sciatica, non-cardiac chest pain, dyspnea, wrist fracture, and neutropenia) were considered unrelated. Three patients died due to disease progression.

Eleven patients across all groups and schedules had at least 1 event considered a dose limiting toxicity (DLT): a treatment-related SAE of Grade 3 febrile neutropenia, a treatment-related SAE of Grade 4 febrile neutropenia, a treatment-related SAE of Grade 4 platelet count decreased, 3 cases of treatment-related SAEs of Grade 4 thrombocytopenia, a treatment-related AE of Grade 4 thrombocytopenia, 3 cases of treatment-related AEs of Grade 4 thrombocytopenia, a treatment-related AE of Grade 4 neutropenia, a treatment-related SAE of Grade 4 neutropenia, a treatment-related AE of Grade 3 diarrhea, 2 cases of treatment-related AEs of Grade 3 nausea, and a treatment related AE of Grade 3 vomiting. Six patients experienced 8 AEs that led to withdrawal from treatment: 1 (Grade 3 AE of cataracts) was considered remotely related to study treatment, 4 (Grade 4 AE of thrombocytopenia/Grade 3 SAE of febrile neutropenia, Grade 2 AE of neutropenia, Grade 3 SAE of febrile neutropenia) were considered possibly related to study treatment, and 3 (Grade 4 SAE of neutropenia, Grade 4 SAE of thrombocytopenia/Grade 4 SAE of neutrophil count decreased) were considered probably related to study treatment.

RG7388 is representative of an entirely new branch of the nutlin family of MDM2 antagonists and the second agent with this mechanism of action sponsored by Roche. As with the lead compound (RO5045337), RG7388 binds selectively to the p53 site on the surface of the MDM2 molecule in vitro with high affinity and can effectively displace p53 from MDM2, leading to stabilization and accumulation of p53 protein and activation of the p53 pathway. RG7388 is from a different chemical series compared to the lead compound and binds with higher potency and selectivity to the MDM2 protein. This follow-on compound has substantially improved pharmacological properties. Preclinical models predict superior efficacy of RG7388 in the clinic at lower doses and exposures. Compared to the lead molecule, lower variability may be seen given that RG7388 does not have significant pH dependent solubility (fasted and fed-state simulated intestinal fluid solubilities are similar). RG7388 at 0.3 μM has equivalent apoptotic activity to RO5045337 at 10-fold higher (3 μM) concentration and at 25 mg/kg has equivalent efficacy to RO5045337 at 4-fold higher dose (100 mg/kg) and better potency when given once weekly.

RG7388 exhibits improved in vitro and in vivo potency against tumor cell lines and xenografts, improved CYP inhibition profile, and 2.5- to 20-fold lower projected human efficacious dose. Preclinical studies have indicated that tumors expressing wild-type p53 may respond to this novel therapeutic strategy that releases p53 from MDM2 inhibition, and tumors with wild-type p53 and MDM2 over-expression or amplification are likely to be the most sensitive. Results from preclinical safety and toxicology studies support further exploration of this compound in cancer patients. In view of the existing unmet medical need in advanced cancers expressing the above molecular signature, RG7388 is believed to be a promising agent that may offer a new therapeutic option.

The use of Pegasys in combination with other targeted agents for the treatment of PV/ET would allow for the administration of lower doses of Pegasys, thereby reducing dose dependent toxicities. Preclinical studies by Lu et al. have demonstrated preferential inhibition of PV CD34+ cell proliferation and colony formation at subtherapeutic doses of Pegasys in combination with Nutlin-3 [33]. Pegasys increases p53 expression through enhanced transcriptional activity via the p38 Map kinase pathway and Nutlin-3 prevents p53 degradation via interruption of the MDM2-p53 interaction [34]. Due to the common downstream target effect of increased tumor suppressor p53 expression with combination Pegasys and Nutlin-3, lower doses of each agent can be used together in PV patients. Thus, the use of RG7388 alone or in combination with Pegasys would be anticipated to enhance p53 expression by different mechanisms and presents a novel approach to the treatment of PV/ET.

ELIGIBILITY:
Inclusion Criteria:

(Patient should meet all the criteria)

* JAK2V617F-positive PV or JAK2V617F-positive ET (confirmed by WHO diagnostic criteria)
* High risk ET/PV [age >60; history of thrombosis] or low risk disease with symptoms [recurrent headaches, paresthesias, pruritus]
* Previously treated with at least one other agent [hydroxyurea, interferon, anagrelide] and determined to be either intolerant/resistant

  -≥18 years of age
* Eastern Cooperative Oncology Group (ECOG) Performance status 0-2
* Acceptable pre-study organ function during screening as defined as: Total bilirubin ≤ 1.5 times the upper limit of normal (ULN) unless due to Gilbert's disease or hemolysis, Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 2.5 times ULN, Serum creatinine ≤ 1.5 x ULN
* Women of childbearing potential and males must agree to use adequate contraception (i.e., hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a female subject become pregnant or suspect she is pregnant while participating in this study, she should inform the treating physician immediately
* Ability to understand and willingness to sign a written informed consent document.

Exclusion Criteria:

* Meets the criteria for post ET/PV MF as defined by the International Working Group-Myeloproliferative Neoplasms Research and Treatment (IWG-MRT)
* Blast phase disease (>20% blasts in the marrow or peripheral blood)
* Acute thrombosis within 3 months of screening
* Uncontrolled intercurrent illness including, but not limited to hepatitis, human immunodeficiency virus (HIV) - positive subjects receiving combination antiretroviral therapy, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, ventricular arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2015-04; Primary Completion 2018-12-19 (Actual); Study Completion 2018-12-19 (Actual)

PRIMARY OUTCOMES:
The dose limiting toxicity of RG7388 | up to 56 days
The dose limiting toxicity of combination of RG7388 and Pegasys | up to 2 years

SECONDARY OUTCOMES:
Hematologic response of PR + CR by modified ELN response criteria | up to 2 years
Molecular response by percent reduction in baseline JAK2V617F allele burden | up to 2 years
Changes in bone marrow histopathologic abnormalities | up to 2 years
Reduction in baseline reticulin/collagen fibrosis | up to 2 years
Incidence of venous and arterial thrombosis | up to 2 years
Changes in MPN related symptoms as measured by the MPN-SAF | up to 2 years

OTHER OUTCOMES:
Pre-treatment wild type P53 status and MDM2 levels as predictors of response to therapy | baseline
Changes in mRNA levels of the following biomarkers : • MIC-1, PCNA, CDKN1A/p21, GDF15, TNFRSF10B/TRAIL-R2, TP53I3/PIG3, and GADD45 | baseline and 2 years
Pre-treatment wild type P53 status and MDM2 levels as predictors of response to combination therapy who failed RG7388 alone and were subsequently treated with combination therapy | baseline

CONTACTS AND LOCATIONS:
Overall Officials: John Mascarenhas, MD, Study Chair — Icahn School of Medicine at Mount Sinai; Ronald Hoffman, MD, Study Chair — Icahn School of Medicine at Mount Sinai
Locations (3):
- United States (3):
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - Wake Forest University Baptist Medical Center, Winston-Salem, North Carolina

REFERENCES:
- [Derived] Mascarenhas J, Lu M, Kosiorek H, Virtgaym E, Xia L, Sandy L, Mesa R, Petersen B, Farnoud N, Najfeld V, Rampal R, Dueck A, Hoffman R. Oral idasanutlin in patients with polycythemia vera. Blood. 2019 Aug 8;134(6):525-533. doi: 10.1182/blood.2018893545. Epub 2019 Jun 5. PMID 31167802